CLINICAL TRIAL: NCT02371707
Title: Interventional, Randomised, Open-label, Two-way Crossover, Single-dose Bioequivalence Study of Idalopirdine in Healthy Subjects Comparing the 60 mg Commercial Tablet (Test) to the 60 mg Clinical Tablet (Reference)
Brief Title: Bioequivalence Study of Idalopirdine Tablets 60 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16052A; 2014-001799-69 (EudraCT Number)
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
MeSH Terms: interventions — (2-(6-fluoro-1H-indol-3-yl)-ethyl)-(3-(2,2,3,3-tetrafluoropropoxy)benzyl)amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Idalopirdine 60 mg formulation A (test) (Experimental)
  Interventions: Drug: Idalopirdine 60 mg formulation A (test)
- Idalopirdine 60 mg formulation B (reference) (Experimental)
  Interventions: Drug: Idalopirdine 60 mg formulation B (reference)

INTERVENTIONS:
Drug: Idalopirdine 60 mg formulation A (test) — Tablet for oral use, single dose
  Other Names: Lu AE58054
  Arms: Idalopirdine 60 mg formulation A (test)
Drug: Idalopirdine 60 mg formulation B (reference) — Tablet for oral use, single dose
  Other Names: Lu AE58054
  Arms: Idalopirdine 60 mg formulation B (reference)

SUMMARY:
This study aims to establish bioequivalence between two tablet formulations of idalopirdine

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women

  -≥18 and ≤55 years of age
* body mass index (BMI) of >18.5 and <30 kg/m2

Exclusion Criteria:

* Pregnant and lactating women

Other protocol defined inclusion and exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Area under the idalopirdine plasma concentration-time curve | 0 to 72 hours post-dose
maximum observed concentration (Cmax) of idalopirdine | 0 to 72 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- Covance, Leeds, United Kingdom